CLINICAL TRIAL: NCT07106476
Title: Effects of Single-Leg Squat Exercises With Different Attentional Focus Techniques on Plantar Pressure Distribution and Posterior Chain Muscle Activation in Individuals With Unilateral Ankle Sprain
Brief Title: Attentional Focus in Single-Leg Squat for Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/08
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Unilateral Ankle Sprain; Chronic Ankle Instability; Muscle Activation; Postural Control; Attentional Focus in Exercise; Neuromuscular Function

STUDY DESIGN:
Intervention Model Description: This study uses a randomized crossover design in which all participants undergo each of the three intervention conditions-internal focus, external focus, and no attentional focus-during the single-leg squat exercise. The order of the conditions is randomized for each participant to reduce sequence and carryover effects. A washout period of 48 hours is maintained between each condition to minimize residual neuromuscular effects. This within-subject design allows for direct comparison of attentional focus strategies on posterior chain muscle activation and plantar pressure parameters.
Who Masked: Outcomes Assessor
Masking Description: Although participants and intervention providers were not masked due to the nature of attentional focus instructions, the outcomes assessor was blinded to the type of attentional focus condition applied during each trial. The assessor responsible for analyzing the sEMG and pedobarographic data was not present during exercise implementation and was unaware of the group assignments. Data files were coded and randomized before analysis to minimize detection bias and ensure objective evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Focus Condition (Experimental): Participants are instructed to focus on their own body movements during the single-leg squat task. Examples of internal focus cues include verbal instructions such as "contract your glutes" or "keep your knee aligned." This condition is designed to direct the participant's attention to specific muscular or joint movements involved in the task.
  Session Length: Each participant completes 3 sets of 8 repetitions on the affected side.
  Rest Period: 1 minute between sets.
  Data Collected: Surface EMG (Gluteus Medius, Biceps Femoris, Lateral Gastrocnemius, Peroneus) and pedobarographic parameters during the movement.
  Interventions: Other: Single-Leg Squat with Internal Focus Intervention
- External Focus Condition (Experimental): Participants are instructed to focus on the effect of the movement in the environment. External cues include statements such as "push against the floor" or "drive your foot downward to move the platform." The goal is to direct attention away from the body and toward the movement outcome.
  Session Length: 3 sets of 8 repetitions on the affected side.
  Rest Period: 1 minute between sets.
  Data Collected: Surface EMG and pedobarographic data.
  Interventions: Other: External Focus Intervention
- No Focus Condition (Experimental): Participants perform the same single-leg squat task without receiving any specific attentional focus instruction. They are simply asked to perform the exercise naturally, as they normally would.
  Session Length: 3 sets of 8 repetitions on the affected side.
  Rest Period: 1 minute between sets.
  Data Collected: Same neuromuscular and plantar pressure data.
  Interventions: Other: No Focus Intervention

INTERVENTIONS:
Other: Single-Leg Squat with Internal Focus Intervention — Administration: Participants were instructed to focus on specific muscular or joint movements during single-leg squats (3 sets of 8 repetitions on the affected side, 1-minute rest between sets). Verbal cues included "contract your glutes" or "keep your knee aligned." Data Collected: Surface EMG (Gluteus Medius, Biceps Femoris, Lateral Gastrocnemius, Peroneus) and pedobarographic parameters.
  Arms: Internal Focus Condition
Other: External Focus Intervention — Administration: Participants were instructed to focus on the environmental effects of single-leg squats (3 sets of 8 repetitions on the affected side, 1-minute rest between sets). Verbal cues included "push against the floor" or "drive your foot downward." Data Collected: Surface EMG (Gluteus Medius, Biceps Femoris, Lateral Gastrocnemius, Peroneus) and pedobarographic parameters.
  Arms: External Focus Condition
Other: No Focus Intervention — Administration: Participants performed single-leg squats naturally without specific attentional instructions (3 sets of 8 repetitions on the affected side, 1-minute rest between sets).
  Data Collected: Surface EMG (Gluteus Medius, Biceps Femoris, Lateral Gastrocnemius, Peroneus) and pedobarographic parameters.
  Arms: No Focus Condition

SUMMARY:
This study investigates the acute effects of single-leg squat exercises conducted under different attentional focus strategies (internal, external, and no focus) on plantar pressure distribution and posterior chain muscle activation in individuals with a history of unilateral ankle sprain. The study aims to determine whether external focus improves neuromuscular efficiency and postural control compared to internal or no attentional focus.

DETAILED DESCRIPTION:
Unilateral ankle sprain is a common condition that compromises proprioception and neuromuscular control, often leading to chronic ankle instability. This randomized crossover trial examines the impact of attentional focus strategies during single-leg squats on surface electromyography (sEMG) activity of posterior chain muscles (gluteus medius, biceps femoris, lateral gastrocnemius, and peroneus) and plantar pressure parameters (COP path length and ellipse area) using pedobarographic analysis. Results may guide rehabilitation protocols by integrating cognitive-motor strategies for improved stability and performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged approximately 18-25 years
* History of unilateral ankle sprain
* Ability to perform single-leg squat exercises
* Willingness to provide written informed consent

Exclusion Criteria:

* Acute musculoskeletal injuries preventing participation
* Neurological or neuromuscular impairments
* Uncorrected visual impairments
* Recent surgery or conditions precluding safe exercise

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Muscle Activation (%MVIC) | Immediately post-intervention in a single session.
  Measured via sEMG for Gluteus Medius, Biceps Femoris, Lateral Gastrocnemius, and Peroneus muscles during single-leg squats under each attentional focus condition.
Center of Pressure (COP) Path Length | Immediately post-intervention in a single session.
  Postural control was assessed immediately after each intervention using a pedobarographic platform. Participants stood barefoot on the affected leg for 30 seconds in a standardized posture (hands on hips, eyes open). The primary outcome in this measure is the COP path length, which represents the total displacement of the pressure center during the trial. Longer COP path lengths indicate greater postural instability.
  Data were sampled at 100 Hz and analyzed using standardized software to evaluate the immediate effects of attentional focus strategies on postural stability.
COP Ellipse Area | Immediately post-intervention, in a single session.
  In the same testing conditions as described above, the COP ellipse area was measured. This reflects the 95% confidence area of sway, providing a spatial measure of postural control. Larger ellipse areas denote impaired balance and increased sway.
  This variable was computed using pedobarographic data sampled at 100 Hz and processed with standardized software.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Fizyoterapi ve Rehabilitasyon Fakültesi, Application Laboratory, Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared publicly due to participant confidentiality and institutional data policy.